CLINICAL TRIAL: NCT04161235
Title: Post-Market Clinical Evaluation of the Zephyr Valve 5.5-LP EBV for Bronchoscopic Lung Volume Reduction (BLVR) Procedures
Brief Title: Post-Market Clinical Evaluation of the Zephyr Valve 5.5-LP EBV
Status: Completed | Type: Observational
Sponsor: Pulmonx Corporation (Industry)
Responsible Party: Sponsor
Other Study IDs: 630-0025-01
Record Dates: First submitted 2019-11-08; First posted 2019-11-13 (Actual); Last update posted 2023-11-15 (Actual); Status verified 2023-11

CONDITIONS: Pulmonary Emphysema
MeSH Terms: conditions — Pulmonary Emphysema

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (1):
- Treatment: Patients undergoing Zephyr Valve treatment with the use of at least one Zephyr Valve 5.5-LP EBV.
  Interventions: Device: The Pulmonx Zephyr Endobronchial Valve (EBV) 5.5- LP

INTERVENTIONS:
Device: The Pulmonx Zephyr Endobronchial Valve (EBV) 5.5- LP — The Zephyr Valves are implantable bronchial valves intended to control airflow in order to improve lung function in patients with hyperinflation associated with severe emphysema and/or to reduce air leaks.

SUMMARY:
This is a Post-Market Evaluation of the Zephyr Valve 5.5-LP EBV to assess Treated Lobar Volume Reduction (TLVR), changes in lung function and the safety profile of the Zephyr Valve treatment with the use of at least one Zephyr Valve 5.5-LP EBV.

DETAILED DESCRIPTION:
This is a multi-center, single-arm, prospective, observational study. Approximately 70 study participants undergoing Zephyr Valve treatment with the use of at least one Zephyr Valve 5.5-LP EBV will be enrolled and followed out to 3 months. Assessments will be conducted at 45 days and 3 months. The evaluation will be conducted at up to 6 sites.

Patients prescribed Zephyr Valve treatment for their emphysema will be consented and will be enrolled only after: 1) determination of little to no collateral ventilation between target and ipsilateral lobes and 2) implantation of at least one Zephyr Valve 5.5-LP EBV. Baseline data will be collected retrospectively after enrollment of a patient in the Post-Market Evaluation. Performance and safety of the Zephyr Valve treatment with the use of at least one Zephyr Valve 5.5-LP will be evaluated post-treatment based on data collected until 3 months after the treatment.

ELIGIBILITY:
Inclusion Criteria:

* Patients with severe emphysema prescribed treatment with Zephyr Valves
* Zephyr Valve Treatment with the use of at least one Zephyr Valve 5.5-LP EBV

Exclusion Criteria:

* Patients determined to have collateral ventilation between the target(s) and ipsilateral lobe(s).
* Patients who undergo Zephyr Valve treatment, but no Zephyr Valve 5.5-LP EBV implanted.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The population evaluated will comprise of patients with hyperinflation associated with severe emphysema that are considered appropriate for the procedure by their physician, confirmed to have little to no collateral ventilation and had at least one Zephyr Valve 5.5-LP EBV implanted during the procedure.
Sampling Method: Non-Probability Sample
Enrollment: 2 (Actual)
Dates: Start 2020-02-05 (Actual); Primary Completion 2021-08-13 (Actual); Study Completion 2021-12-30 (Actual)

PRIMARY OUTCOMES:
Treated Lobar Volume Reduction (TLVR) responders | 45 days
  The percentage of patients treated with the Zephyr Valve 5.5-LP EBV who achieved a Treated Lobar Volume Reduction (TLVR) of the treated lobe (s) of ≥350ml as seen via HRCT at 45-days.

OTHER OUTCOMES:
Treated Lobar Volume Reduction (TLVR) changes from Baseline | 45 days
  Treated Lobar Volume Reduction (TLVR) as seen via HRCT at 45-days (absolute and percent changes from baseline).
Lobar occlusion | 45 days
  Lobar occlusion of the treated lobe at 45-days post-procedure as visualized by HRCT.
Post-Bronchodilator Forced Expiratory Volume in 1 second (FEV1) | 3 months
  Post-Bronchodilator Forced Expiratory Volume in 1 second (FEV1) at 3-months (absolute and percent changes from baseline).
Residual Volume (RV) | 3 months
  Residual Volume at 3 months, when available (absolute and percent changes from baseline).
Total Lung Capacity | 3 months
  Total Lung Capacity (TLC) at 3 months, when available (absolute and percent changes from baseline).
Inspiratory Capacity | 3 months
  Inspiratory Capacity (IC) at 3 months, when available (absolute and percent changes from baseline).
Residual Volume/Total Lung Capacity (RV/TLC) | 3 months
  RV/TLC ratio at 3 months, when available (absolute and percent changes from baseline).
Inspiratory Capacity/Total Lung Capacity (IC/TLC) | 3 months
  IC/TLC ratio at 3 months, when available (absolute and percent changes from baseline).

CONTACTS AND LOCATIONS:
Locations (3):
- Ruhrlandklinik Essen - Universitätsmedizin, Essen, Germany
- University Hospital of Zurich, Zurich, Switzerland
- Royal Brompton Hospital, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No